CLINICAL TRIAL: NCT04935827
Title: Seasonal Differences in Home Dialysis Uptake and Initiating Dialysis in the Hospital
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eugene Lin, Assistant Professor, University of Southern California
Other Study IDs: HS-18-00530-2; K08DK118213 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Dialysis; Peritoneal Dialysis; Hospitalizations
MeSH Terms: interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients initiating dialysis for end-stage kidney disease: Patients whose start of dialysis is from 12/1/2007-11/30/2017. We use the following inclusion criteria:
  * Adult (>= 18 years old)
  * Did not die or have a transplant prior to the 90th day of dialysis
  * Valid medical evidence form
  * Medicare Part A/B as primary payer in the 30 days prior to initiating dialysis
  * Initiating dialysis in the USA
  Interventions: Other: Season of Year; Other: Hospitalized 14 days prior to dialysis

INTERVENTIONS:
Other: Season of Year — We stratify patients into 4 groups based on the season of the year (between 12/1/2007-11/30/2017)
  * Winter: December, January, February
  * Spring: March, April, May
  * Summer: June, July, August
  * Fall: September, October, November
Other: Hospitalized 14 days prior to dialysis — We further stratify patients into 3 groups based on whether they were hospitalized within 14 days prior to dialysis
  * Group 1: No hospitalization prior to dialysis
  * Group 2: Hospitalized within 14 days prior to dialysis for an acute infectious respiratory condition or one of the following acute cardiac conditions (arrhythmia, myocardial infarction, stroke, or fluid overload)
  * Group 3: Hospitalized within 14 days prior to dialysis for a condition not in Group 2

SUMMARY:
This study will investigate whether home dialysis uptake varies by the season of year. We will also investigate whether hospitalizations around the time of dialysis also vary by season of year and whether hospitalizations are associated with reduced home dialysis starts and sustained home dialysis uptake.

ELIGIBILITY:
Inclusion Criteria:

* Started dialysis in the USA for end-stage kidney disease from 12/1/2007-11/30/2017
* No transplant or death prior to day 90 of dialysis
* Medicare Parts A/B as primary payer 30 days prior to starting dialysis
* Valid Medicare Evidence Form (Form 2728)

Exclusion Criteria:

* As above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults with fee-for-service Medicare coverage initiating dialysis for end-stage kidney disease in the United States from 12/1/2007-11/30/2017
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Type of dialysis modality at the start of dialysis | Day 1 of dialysis
  Whether patient started with home dialysis or in-center dialysis at the start of dialysis
Type of dialysis modality at the end of month 3 of dialysis | End of month 3 of dialysis
  Whether patient was using home dialysis or in-center dialysis at the end of month 3 of dialysis (day 84)
Type of dialysis modality at the end of month 6 of dialysis | End of month 6 of dialysis
  Whether patient was using home dialysis or in-center dialysis at the end of month 6 of dialysis (day 168)
Type of dialysis modality at the end of month 9 of dialysis | End of month 9 of dialysis
  Whether patient was using home dialysis or in-center dialysis at the end of month 9 of dialysis (day 252)
Type of dialysis modality at the end of month 12 of dialysis | End of month 12 of dialysis
  Whether patient was using home dialysis or in-center dialysis at the end of month 12 of dialysis (day 336)
Mortality in the first year | 1 year of dialysis
  Whether the patient died in the first year of dialysis and the number of days the patient survived
  - Censored for transplantation, loss to follow-up

IPD SHARING:
Plan to Share IPD: No
Data are protected by a DUA from the United States Renal Data System. Researchers interested in obtaining the data must obtain a DUA. We will share programs to generate the analyses via an open source sharing resource.

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04935827/SAP_000.pdf